CLINICAL TRIAL: NCT03028714
Title: The Impact of an Educational Intervention on Nutrition Knowledge, Dietary Habits, BMI and Physical Activity, in University Students in the United Kingdom (UK).
Brief Title: The Impact of Online Quiz-games on Nutrition Knowledge and Related Outcomes Among University Students.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kingston University (Other)
Collaborators: St George's, University of London (Other); King's College London (Other)
Responsible Party: Principal Investigator, Katerina Belogianni, Principal Investigator, Kingston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FREC 2016-04-001
Record Dates: First submitted 2017-01-16; First posted 2017-01-23 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: University; College; University students; Health education; Educational techonology; Internet; Nutrition knowledge; Eating behaviour; Diet; Physical Activity; Weight gain prevention
MeSH Terms: conditions — Behavior; Health Education; Feeding Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-based nutrition education (Experimental): Participants will receive access to a website including educational information about nutrition and related topics. Through the website they will be asked to play online quiz-games relevant to the content of the website to improve their knowledge.
  Interventions: Behavioral: Technology-based nutrition education
- Control group (No Intervention): Participants in the control group will receive no intervention.

INTERVENTIONS:
Behavioral: Technology-based nutrition education — All participants will undertake anthropometric measurements and assessments of blood pressure and blood glucose. They will be also asked to complete online questionnaires with regards to nutrition and physical activity. Participants in the intervention group will receive additional access to a website, providing information about nutrition topics including alcohol and physical activity. Through the website participants will be asked to play online quiz-games related to the nutrition topics. Each play will include game elements such as time, point collection and graphics. Participants will be asked to play the games as much as they want to improve their scores and to use the website as a reference tool.
  Arms: Technology-based nutrition education

SUMMARY:
Metabolic risk factors, such as central obesity, increase the risk of chronic diseases in adulthood and are prevalent in many university students. Increasing the knowledge about healthy nutrition and physical activity can positively impact students' lifestyle and prevent weight gain. This study aims to investigate the impact of online educational methods on nutrition knowledge, dietary habits, BMI, and physical activity in a sample of university students in the UK. Anthropometric measurements will be assessed and questionnaires will be completed at the beginning and at the end of the study. Written consent will be sought, the voluntary nature of participation will be emphasized while anonymity and confidentiality will be strictly maintained.

DETAILED DESCRIPTION:
The intervention is a randomized-controlled trial with two data collection points: one at the beginning and one at the end of the study. The study will include healthy students from two UK Universities, who they will be randomly assigned either to the intervention or to the control group. Participants in both groups will be asked to undertake measurements and complete questionnaires before and after the study. Measurements include the assessment of BMI, body fat, lean mass, waist-to-hip ratio, systolic and diastolic blood pressure and blood glucose. In addition, nutrition knowledge and dietary habits will be estimated using online questionnaires as well as the level of physical activity using the IPAQ questionnaire and pedometers. Participants in the intervention group will receive access to an educational website including information about fruit and vegetables, fat, sugars, fast-food, meat, salt, meals and snacks, food labels, exercise, and alcohol. Each category will be linked to an online quiz-game that will include questions related to the topic. Students will be asked to play the games as much as they want to improve their knowledge scores. Access to the website and the games will be available for 10 weeks. Participants in the control group will receive no intervention. After 10 weeks, participants will be asked to undertake the same measurements and complete the same questionnaires as they did in the beginning of the study. The study aims to investigate the effectiveness of an online educational intervention, using game elements, on the level of nutrition knowledge of students, as well as, whether any changes in knowledge impact changes in dietary habits, physical activity and weight-related factors.

ELIGIBILITY:
Inclusion Criteria:

* Currently studying at Kingston University, London or at St George's, University of London, as an undergraduate or postgraduate student or undertaking research within one of the two organizations.
* Aged between 18 and 34 years.
* Generally, in good health.

Exclusion Criteria:

* Not currently studying at Kingston University, London or at St George's, University of London.
* Less than 18 or more than 34 years old.
* Suffering a long-term disease or condition that requires a special treatment or diet.
* Suffering a mobility impairment or injury that doesn't allow undertaking moderate physical activity.
* Pregnant or breast-feeding.

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Level of nutrition knowledge (score in units) | One year
  The level of nutrition knowledge will be assessed using the General Nutrition Knowledge Questionnaire (GNKQ) (Kliemann et al., 2016). The GNKQ includes questions with multiple choice answers, presented in 4 sections: section 1 is related to dietary recommendations, section 2 is related to food groups, section 3 is related to health food choices and section 4 is related to diet, disease and weight association. Each correct answer gets a point (otherwise null) and the maximum score is 88 for the overall questionnaire, 18 for section 1, 36 for section 2, 13 for section 3 and 21 for section 4.

SECONDARY OUTCOMES:
Dietary habits (score in units) | One year
  Dietary habits will be assessed using the questionnaire of Leppälä, J. et al. (2010). The questionnaire includes 18 questions in relation to whole grain products, fat containing foods, dairy products, vegetables and fruits, sugar and meal pattern. A scoring system is provided as a manual to calculate the total score based on the answer given to each question. The total score represents diet quality (Index of Diet Quality) and can be ranged from 0-15, with 9 or less points indicating a poor diet quality.
Physical activity [vigorous activity (days/week, minutes/week), moderate activity (days/week, minutes/week), walking (days/week, minutes/week), sitting time (minutes/week)]. | One year
  Physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ-short) (Craig et al., 2003). The questionnaire includes questions regarding 1) days per week and time (minutes) spent on one of those days doing vigorous activity, 2) days per week and time (minutes) spent on one of those days doing moderate activity, 3) days per week and time (minutes) spent on one of those days walking and 4) time (minutes) spent the last week sitting on a week day.
Physical activity (number of steps/week). | One year
  Pedometers will be used to calculate the amount of physical activity by counting daily number of steps.
Body Mass Index (BMI) (kg/m2) | 1 year
  BMI (kg/m2) will be estimated after measuring body weight (kg), using an analog scale and height (in meters), using a stadiometer.
Body fat (%) | 1 year
  Body fat (%) will be estimated using a TANITA body fat analyzer.
Lean mass (kg) | 1 year
  Lean mass (kg) will be estimated using a TANITA body fat analyzer.
Waist-to-hip ratio (WHR) | 1 year
  To calculate waist-to-hip ratio a measuring tape will be used to measure waist circumference (cm) and hip circumference (cm) separately. Waist circumference (cm) will be measured at the midpoint between the top of the iliac crest and the lower margin of the last palpable rib in the mid axillary line. Hip circumference (cm) will be measured at the largest circumference of the buttocks.
Blood pressure (mmHg) | 1 year
  Systolic (mmHg) and diastolic (mmHg) blood pressure will be measured using an electronic sphygmomanometer. The participant will be in a relaxed, quiet room at a comfortable temperature and a short period of 5 minutes rest will precede the measurement.The measurement will be undertaken twice.
Blood glucose (mmol/l) | 1 year
  Blood glucose levels (mmol/l) will be measured by finger pricking using a blood glucose meter. The participant will be asked to be fasted.

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Belogianni, PhD, Principal Investigator — Kingston University, London
Locations (1):
- Kingston University, London & St George's, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kliemann N, Wardle J, Johnson F, Croker H. Reliability and validity of a revised version of the General Nutrition Knowledge Questionnaire. Eur J Clin Nutr. 2016 Oct;70(10):1174-1180. doi: 10.1038/ejcn.2016.87. Epub 2016 Jun 1. PMID 27245211
- [Result] Leppala J, Lagstrom H, Kaljonen A, Laitinen K. Construction and evaluation of a self-contained index for assessment of diet quality. Scand J Public Health. 2010 Dec;38(8):794-802. doi: 10.1177/1403494810382476. Epub 2010 Sep 16. PMID 20846997
- [Result] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694